CLINICAL TRIAL: NCT05087628
Title: Phase 2a, Randomized, Double-blind, Placebo-controlled Trial of PRV-3279 EVAluation In Lupus
Brief Title: PRV-3279-2a Trial in Systemic Lupus
Acronym: PREVAIL-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: termination for strategy reasons
Sponsor: Provention Bio, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-3279-2a; ACT18113 (Other: Sanofi Identifier)
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRV-3279 (Experimental): Sterile solution for intravenous administration, every 4 weeks
  Interventions: Biological: PRV-3279
- Placebo (Experimental): Sterile solution for intravenous administration, every 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PRV-3279 — Bi-specific antibody-based molecule
  Other Names: SAR446811
  Arms: PRV-3279
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The PREVAIL-2 study is designed to assess the safety and potential efficacy of PRV-3279 in flare prevention in systemic lupus erythematosus (SLE) patients with active disease after amelioration induced by corticosteroid treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study in adult patients with active SLE. Approximately 100 eligible patients will be randomized at a 1:1 ratio to receive treatment with either PRV-3279 or placebo.

Eligible subjects include male or female adults, 18 to 70 years of age, with a diagnosis of SLE for at least 6 months.

The study drug will be administered every 4 weeks for 20 weeks in a double-blind fashion, followed by an 8-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of SLE for at least 6 months prior to the Screening visit
2. Meet the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) criteria for SLE at Screening
3. Have moderate to severe disease activity despite stable standard-of-care medication defined as:

   At screening: hSLEDAI score ≥6 (≥4 points of which must come from non-serological finding), OR at least one BILAG A or one B score; At randomization: ≥4-point drop in hSLEDAI, OR one BILAG letter grade improvement in at least one A or B score present at Screening, and investigator or central adjudication committee (CAC) rating of definite improvement or major or complete improvement
4. Able and willing to stop all lupus treatments, except antimalarials, corticosteroids (prednisone equivalent ≤ 10 mg), and NSAIDs

Exclusion Criteria:

1. Active lupus nephritis or active central nervous system manifestations of SLE
2. Other inflammatory or autoimmune diseases that, in the opinion of the Investigator or CAC, may confound efficacy evaluations
3. Common variable immunodeficiency syndrome or any other clinically significant immunodeficiency
4. Known COVID-19 infection in the 4 weeks before Screening or positive SARS-CoV-2 RNA test
5. Received a live attenuated vaccine within 2 months of Screening, received a non-live or mRNA vaccine within 2 weeks of Screening, or expecting to receive any vaccine during the study period
6. Any recent infection requiring antibiotics within two weeks of Screening or any recent infection requiring IV antibiotics or hospitalization within 1 month of Screening
7. Any condition for which, in the opinion of the Investigator or CAC, participation in the study would not be in the best interest of the patient (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments
8. Participated in any interventional clinical trial within 42 days prior to Screening or within five half-lives of the investigational product, whichever is longer
9. Received rituximab or equivalent treatment that depletes B cells within 6 months of Screening unless return of B cells to pre-treatment value or normal range can be demonstrated.
10. Received tumor necrosis factor inhibitors, interleukin antagonists, or other biologics, including belimumab, within 42 days or five half-lives of the agent, whichever is longer.
11. Received IV immunoglobulin (IVIG) or IV cyclophosphamide within 2 months, prednisone ≥ 100 mg/day for more than 30 days within 2 months, or plasmapheresis within two months of the Screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of PRV-3279 to prevent flare, defined by LFA international consensus definition of flare, worsening on CGIC, and increase in hSLEDAI/BILAG scores | 24 weeks
  A flare is defined according to LFA international consensus definition of flare, worsening on Clinician's Global Impression of Change (CGIC), increases in hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI)/British Isles Lupus Assessment Group (BILAG) Index scores

SECONDARY OUTCOMES:
To evaluate whether PRV-3279 prolongs the duration of disease amelioration induced by corticosteroids | 24 weeks
  Time to treatment failure
To evaluate the safety of PRV-3279 | 32 weeks
  Frequency of TEAEs, SAEs, TEAEs leading to drug withdrawal, AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (36):
- United States (22):
  - Medvin Clinical Research - Apple Valley- Site Number : 133, Apple Valley, California
  - Medvin Clinical Research - Covina - West San Bernardino Road- Site Number : 106, Covina, California
  - University of California San Diego - La Jolla- Site Number : 108, La Jolla, California
  - University of California Los Angeles Medical Center- Site Number : 122, Los Angeles, California
  - Facey Medical Group - Los Angeles- Site Number : 126, Los Angeles, California
  - Desert Medical Advances- Site Number : 114, Rancho Mirage, California
  - Medvin Clinical Research - Tujunga- Site Number : 119, Tujunga, California
  - Medvin Clinical Research - Whittier- Site Number : 118, Whittier, California
  - Highlands Advanced Rheumatology & Arthritis Center- Site Number : 116, Avon Park, Florida
  - Center for Rheumatology, Immunology and Arthritis- Site Number : 109, Fort Lauderdale, Florida
  - Millennium Research- Site Number : 111, Ormond Beach, Florida
  - D&H Tamarac Research Center- Site Number : 123, Tamarac, Florida
  - Florida Hospital Tampa- Site Number : 107, Tampa, Florida
  - Vernon Hills Medical Associates- Site Number : 128, Vernon Hills, Illinois
  - Ochsner Medical Center - Jefferson Highway- Site Number : 113, New Orleans, Louisiana
  - Revival Research Corporation - Michigan - ClinEdge - PPDS- Site Number : 124, Troy, Michigan
  - University of Toledo Medical Center- Site Number : 110, Toledo, Ohio
  - Yale University School of Medicine- Site Number : 125, Pittsburgh, Pennsylvania
  - Grapevine Rheumatology Clinic- Site Number : 103, Grapevine, Texas
  - Accurate Clinical Management - Greenhouse Road- Site Number : 104, Houston, Texas
  - Accurate Clinical Research - Houston Resource Parkway- Site Number : 105, Houston, Texas
  - Sun Research Institute- Site Number : 121, San Antonio, Texas
- China (9):
  - Investigational Site Number : 310, Beijing
  - Investigational Site Number : 301, Beijing
  - Investigational Site Number : 309, Changchun
  - Investigational Site Number : 302, Guangzhou
  - Investigational Site Number : 303, Nanchang
  - Investigational Site Number : 307, Nanjing
  - Investigational Site Number : 306, Shanghai
  - Investigational Site Number : 305, Tianjin
  - Investigational Site Number : 304, Wuhan
- Hong Kong (2):
  - Investigational Site Number : 202, Pok Fu Lam
  - Investigational Site Number : 201, Tuenmen
- Puerto Rico (3):
  - Centro Reumatologico de Caguas- Site Number : 112, Caguas
  - Private Practice - Dr. Karina Vila Rivera- Site Number : 117, San Juan
  - BCR Medical Center Inc.- Site Number : 129, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org